CLINICAL TRIAL: NCT00363545
Title: A Study to Assess the Immunogenicity, Reactogenicity and Safety of 2 Different Formulations of GSK Biologicals' Live Attenuated HRV Vaccine, Given as a Two-dose Primary Vaccination, in Healthy Infants Previously Uninfected With HRV
Brief Title: To Assess Immunogenicity, Reactogenicity & Safety of 2 Formulations of GSK's HRV Vaccine as 2-dose Vaccination (Infants)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 107077
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Infections, Rotavirus
Keywords: Prophylaxis against gastroenteritis caused by Rotavirus
MeSH Terms: conditions — Rotavirus Infections

ARMS (2):
- Liquid Rotarix Group (Experimental): Healthy male and female infants, between and including 6-12 weeks of age, who received two oral doses of the liquid formulation of the Rotarix™ vaccine, according to a 0, 2 month schedule.
  Interventions: Biological: Liquid formulation of HRV vaccine
- Lyophilized Rotarix Group (Experimental): Healthy male and female infants, between and including 6-12 weeks of age, who received two oral doses of the lyophilized formulation of the Rotarix™ vaccine, according to a 0, 2 month schedule.
  Interventions: Biological: Lyophilized formulation of HRV vaccine

INTERVENTIONS:
Biological: Lyophilized formulation of HRV vaccine — Lyophilized formulation of HRV vaccine
  Arms: Lyophilized Rotarix Group
Biological: Liquid formulation of HRV vaccine — Liquid formulation of HRV vaccine
  Arms: Liquid Rotarix Group

SUMMARY:
This trial will be conducted to evaluate the immunogenicity, reactogenicity and safety of the liquid formulation of GSK Biologicals' HRV vaccine compared to the lyophilized formulation of GSK Biologicals' HRV vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infant between, and including, 6 and 12 weeks of age born after a gestation period of 36 to 42 weeks.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* se of any investigational or non-registered product (drug or vaccine) other than the HRV vaccine within 30 days preceding the first dose of HRV vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccines not foreseen by the study protocol except for DTPw, HBV/Hib and OPV vaccines within 14 days before each dose of HRV vaccine and ending 14 days after.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Household contact with an immunosuppressed individual or pregnant women.
* Previous confirmed occurrence of RV GE.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1274 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2007-04-12 (Actual); Study Completion 2007-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Panama (3):
  - GSK Investigational Site, David
  - GSK Investigational Site, La Chorrera
  - GSK Investigational Site, Panama City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Velasquez AA et al. Immunogenicity of The Oral Live Attenuated Human Rotavirus Vaccine RIX4414 (Rotarix™) Oral Suspension (Liquid Formulation) Co-administered with Childhood Vaccinations in Panama. Poster presented at the 13th International Congress on Infectious Diseases (ICID), Kuala Lumpur, Malaysia, 19-22 June 2008.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 107077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Started | 636 | 638
Completed | 592 | 581
Not Completed | 44 | 57
Not completed — Serious Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 12 | 15
Not completed — Migrated/moved from study area | 3 | 6
Not completed — Lost to follow-up (incompl. vaccination) | 14 | 18
Not completed — Lost to follow-up (complete vaccination) | 14 | 17
Not completed — Others | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group | Total
Number analyzed (Participants) | 636 | 638 | 1274
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.6 (0.87) | 8.6 (0.86) | 8.6 (0.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 294 | 316 | 610
  Male | 342 | 322 | 664

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against Human Rotavirus
Description: A seroconverted subject was defined as a vaccinated subject who had an anti-rotavirus IgA antibody concentration equal to or above (≥) 20 units per milliliter (U/mL) and who was initially (i.e. prior to the first dose of Rotarix™ vaccine) negative for rotavirus.
Time Frame: At 1 to 2 months after the second vaccine dose (Months 3-4)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available at post-sampling time point.
Measure: Number; unit: Subjects
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Number analyzed (Participants) | 449 | 434
Subjects | 363 | 319

2. Secondary Outcome: Concentrations of Anti-rotavirus IgA Antibodies
Description: Anti-rotavirus IgA antibody concentrations assessed by using the Enzyme-Linked Immunosorbent Assay (ELISA) are presented as geometric mean concentrations (GMCs), expressed in units per milliliter (U/mL).
Time Frame: At 1 to 2 months after the second vaccine dose (Months 3-4)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data were available at post-sampling time point.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Number analyzed (Participants) | 449 | 434
U/mL | 151.2 [128.0 to 178.7] | 111.7 [93.5 to 133.4]

3. Secondary Outcome: Number of Subjects With Vaccine Take for Anti-rotavirus IgA Antibodies
Description: Vaccine take was defined as appearance of serum anti-rotavirus IgA antibodies in post-vaccination sera at a concentration of ≥ 20 U/mL and/or vaccine virus excretion in any stool sample collected from Day 0 to Month 4, for subjects initially negative for rotavirus. The analysis was performed on the stool analysis subset, which included 100 subjects per group.
Time Frame: At 1 to 2 months after the second vaccine dose (Months 3-4)
Population: The analysis was performed on the ATP cohort for immunogenicity stool analysis subset, defined as the first 200 subjects for whom pre-vaccination stool samples were available and with available anti-rotavirus IgA antibody results at post sampling time point or with vaccine virus in stools collected after the first vaccine dose up to Month 4.
Measure: Number; unit: Subjects
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Number analyzed (Participants) | 81 | 71
Subjects | 67 | 51

4. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were cough/runny nose, diarrhea, fever [defined as rectal temperature equal to or above 38 degrees Celsius (°C)], irritability/fussiness (Irr./Fuss.), loss of appetite and vomiting. Any = occurrence of the symptom regardless of intensity grade. Grade 3 cough/runny nose = cough/runny nose that prevented normal activity. Grade 3 diarrhea = 6 or more than (≥) 6 looser than normal stools/day. Grade 3 irritability/fussiness (Irr./Fuss.) = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 vomiting = 3 or more than (≥) 3 episodes of vomiting/day. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 15-day (Day 0-14) follow-up period, after each vaccine dose and across doses, up to 4 months.
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one study vaccine administration documented and with symptoms sheet filled in.
Measure: Number; unit: Subjects
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Number analyzed (Participants) | 636 | 638
Subjects
  Any Cough/runny nose, Dose 1 | 234 | 252
  Grade 3 Cough/runny nose, Dose 1 | 22 | 20
  Related Cough/runny nose, Dose 1 | 31 | 22
  Any Diarrhea, Dose 1 | 43 | 34
  Grade 3 Diarrhea, Dose 1 | 8 | 11
  Related Diarrhea, Dose 1 | 19 | 14
  Any Fever (Rectal), Dose 1 | 296 | 292
  Grade 3 Fever (Rectal), Dose 1 | 12 | 12
  Related Fever (Rectal), Dose 1 | 148 | 161
  Any Irr./Fuss., Dose 1 | 343 | 352
  Grade 3 Irr./Fuss., Dose 1 | 35 | 35
  Related Irr./Fuss., Dose 1 | 150 | 156
  Any Loss of appetite, Dose 1 | 152 | 163
  Grade 3 Loss of appetite, Dose 1 | 8 | 6
  Related Loss of appetite, Dose 1 | 48 | 55
  Any Vomiting, Dose 1 | 131 | 129
  Grade 3 Vomiting, Dose 1 | 36 | 27
  Related Vomiting, Dose 1 | 24 | 20
  Any Cough/runny nose, Dose 2: number analyzed (Participants) | 605 | 597
  Any Cough/runny nose, Dose 2 | 239 | 239
  Grade 3 Cough/runny nose, Dose 2: number analyzed (Participants) | 605 | 597
  Grade 3 Cough/runny nose, Dose 2 | 19 | 23
  Related Cough/runny nose, Dose 2: number analyzed (Participants) | 605 | 597
  Related Cough/runny nose, Dose 2 | 31 | 42
  Any Diarrhea, Dose 2: number analyzed (Participants) | 605 | 597
  Any Diarrhea, Dose 2 | 23 | 27
  Grade 3 Diarrhea, Dose 2: number analyzed (Participants) | 605 | 597
  Grade 3 Diarrhea, Dose 2 | 5 | 9
  Related Diarrhea, Dose 2: number analyzed (Participants) | 605 | 597
  Related Diarrhea, Dose 2 | 7 | 5
  Any Fever (Rectal), Dose 2: number analyzed (Participants) | 605 | 597
  Any Fever (Rectal), Dose 2 | 283 | 274
  Grade 3 Fever (Rectal), Dose 2: number analyzed (Participants) | 605 | 597
  Grade 3 Fever (Rectal), Dose 2 | 23 | 14
  Related Fever (Rectal), Dose 2: number analyzed (Participants) | 605 | 597
  Related Fever (Rectal), Dose 2 | 139 | 148
  Any Irr./Fuss., Dose 2: number analyzed (Participants) | 605 | 597
  Any Irr./Fuss., Dose 2 | 280 | 298
  Grade 3 Irr./Fuss., Dose 2: number analyzed (Participants) | 605 | 597
  Grade 3 Irr./Fuss., Dose 2 | 31 | 23
  Related Irr./Fuss., Dose 2: number analyzed (Participants) | 605 | 597
  Related Irr./Fuss., Dose 2 | 137 | 155
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 605 | 597
  Any Loss of appetite, Dose 2 | 136 | 138
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 605 | 597
  Grade 3 Loss of appetite, Dose 2 | 8 | 6
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 605 | 597
  Related Loss of appetite, Dose 2 | 45 | 61
  Any Vomiting, Dose 2: number analyzed (Participants) | 605 | 597
  Any Vomiting, Dose 2 | 85 | 82
  Grade 3 Vomiting, Dose 2: number analyzed (Participants) | 605 | 597
  Grade 3 Vomiting, Dose 2 | 20 | 22
  Related Vomiting, Dose 2: number analyzed (Participants) | 605 | 597
  Related Vomiting, Dose 2 | 5 | 7
  Any Cough/runny nose, Across doses | 335 | 342
  Grade 3 Cough/runny nose, Across doses | 36 | 41
  Related Cough/runny nose, Across doses | 56 | 58
  Any Diarrhea, Across doses | 61 | 59
  Grade 3 Diarrhea, Across doses | 13 | 20
  Related Diarrhea, Across doses | 24 | 19
  Any Fever (Rectal), Across doses | 405 | 406
  Grade 3 Fever (Rectal), Across doses | 34 | 26
  Related Fever (Rectal), Across doses | 220 | 240
  Any Irr./Fuss., Across doses | 401 | 427
  Grade 3 Irr./Fuss., Across doses | 55 | 49
  Related Irr./Fuss., Across doses | 211 | 238
  Any Loss of appetite, Across doses | 218 | 234
  Grade 3 Loss of appetite, Across doses | 16 | 11
  Related Loss of appetite, Across doses | 83 | 95
  Any Vomiting, Across doses | 162 | 167
  Grade 3 Vomiting, Across doses | 44 | 43
  Related Vomiting, Across doses | 29 | 26

5. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days after any vaccine dose (Day 0-30) post-vaccination, up to 4 months
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one study vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Number analyzed (Participants) | 636 | 638
Subjects | 276 | 285

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the entire study period (from Day 0 to Month 4)
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Number analyzed (Participants) | 636 | 638
Subjects | 37 | 38

7. Secondary Outcome: Number of Subjects With Rotavirus in Stool Samples Collected During Gastroenteritis Episodes
Description: The number of subjects with rotavirus (vaccine strain or wild-type rotavirus) in stool samples collected during gastroenteritis episodes from the first dose (Dose 1) of Rotarix™ vaccine up to Visit 3, as follows: between Dose 1 and before Dose 2, between Dose 2 and Visit 3 and between Dose 1 and Visit 3.
Time Frame: From the first vaccine dose (Dose 1) up to Month 4
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Number analyzed (Participants) | 636 | 638
Subjects
  Dose 1-Dose 2 (N=636;638) | 4 | 2
  Dose 2-Visit 3 (N=605;597) | 1 | 0
  Dose 1-Visit 3 (N=636;638) | 5 | 2

ADVERSE EVENTS:
Time Frame: Solicited general symptoms: within the 15-day (Day 0-14) follow-up period after each vaccine dose; Unsolicited AEs: within 31 days (Day 0-30) after any vaccine dose; SAEs: throughout the entire study period (from Day 0 to Month 4).
Arm/Group | Liquid Rotarix Group | Lyophilized Rotarix Group
Serious Adverse Events (participants affected / at risk) | 37/636 | 38/638
Other Adverse Events (participants affected / at risk) | 553/636 | 556/638
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid Rotarix Group (N=636) | Lyophilized Rotarix Group (N=638)
Bronchiolitis (Infections and infestations) | 22 | 20
Pneumonia (Infections and infestations) | 10 | 7
Gastroenteritis (Infections and infestations) | 4 | 6
Bronchopneumonia (Infections and infestations) | 3 | 4
Gastro esophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Hypoxic encephalopathy (Nervous system disorders) | 1 | 0
Infantile spasms (Nervous system disorders) | 1 | 0
Milk allergy (Immune system disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Omphalitis (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Liquid Rotarix Group (N=636) | Lyophilized Rotarix Group (N=638)
Cough/runny nose (General disorders) | 335 | 342
Diarrhea (General disorders) | 61 | 59
Fever (Rectal) (General disorders) | 405 | 406
Irritability/ Fussiness (General disorders) | 401 | 427
Loss of appetite (General disorders) | 218 | 234
Vomiting (General disorders) | 162 | 167
Nasopharyngitis (Infections and infestations) | 164 | 162
Bronchiolitis (Infections and infestations) | 38 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.